CLINICAL TRIAL: NCT03233620
Title: Effectiveness of Contemporary Knee Arthroplasty in Working-age Patients: a Prospective Study With 2-year Follow-up
Brief Title: Effectiveness of Contemporary Knee Arthroplasty in Working-age Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coxa, Hospital for Joint Replacement (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R11178
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Knee Osteoarthritis
Keywords: knee arthroplasty; working-age; patient related outcome measures
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- working age patients (Other): Prospective cohort of 250 patients.
  Interventions: Other: Knee arthroplasty

INTERVENTIONS:
Other: Knee arthroplasty — Effectiveness of knee arthroplasty surgery.

SUMMARY:
The aim of our study was to assess the effectiveness of contemporary knee arthroplasty in working-age patients (< 65 years) by conducting a prospective cohort study with 2-year follow up. Outcomes were measured comprehensively using various patient-reported outcome measures (PROMs) to provide information on the effect of knee arthroplasty on pain, satisfaction, physical activity, activities of daily living, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or less and
* Scheduled for either TKA or unicondylar knee arthroplasty (UKA)

Exclusion Criteria:

* rheumatoid arthritis or other inflammatory diseases
* unwilling to provide informed consent
* physical, mental, or neurological conditions that could comprise the patient´s ability and compliance with postoperative rehabilitation and follow-up (e.g., drug or alcohol abuse, serious mental illness, general neurological conditions such as Parkinson's disease, multiple sclerosis (MS), etc.)
* known sensitivity to materials in the devices.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of contemporary knee arthroplasty in working-age patients | 2 years
  PROMs

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leppanen S, Niemelainen M, Huhtala H, Eskelinen A. Mild knee osteoarthritis predicts dissatisfaction after total knee arthroplasty: a prospective study of 186 patients aged 65 years or less with 2-year follow-up. BMC Musculoskelet Disord. 2021 Aug 5;22(1):657. doi: 10.1186/s12891-021-04543-8. PMID 34353317